CLINICAL TRIAL: NCT06230627
Title: University of Mosul, College of Physical Education and Sport Sciences & University of Sfax, High Institute of Sport and Physical Education at Sfax
Brief Title: Feasibility of Home-Based Rehabilitation on Body Composition, Some Anthropometric Measures and Muscular Strength After Interruption 4-5 Years of Spinal Cord Injury: Serial Cases Study on ISIS War Survivors in Iraq
Acronym: HBRP-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mosul (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Mosul
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Rehabilitation; Exercises
Keywords: Spinal Cord Injury, Anthropometric, Muscles Strength, Tele-rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Eternal Intervention (Home-Based Rehabilitation Program) Three groups :
  Experimental group with SCI + Control group 1 with SCI + Control group 2 Healthy people
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: There were two control groups in this study, the first were people with SCI who only conducted the pre-post1 and post2-tests, additionally, the second group were healthy people also they just conducted the pre-post1 and post2-tests. The authors used these groups to control the changes which may happen with time which could affect the results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rehabilitation program (Experimental): The Home-Based Rehabilitation Program (HBRP) As a first procedure, detailed interviews were conducted with each participant at the beginning of the study to gather information about their physical, psychological, and social well-being. This information helped the authors create personalized rehabilitation plans for each participant to ensure their participation in the study for the entire 6 months period. Through our study objectives, the authors used body composition such as height, weight, BMI and some anthropometric measurements for body parts circumferences by using tape measurements. Also, muscle strength tests were performed on participants' lower and upper extremities, head, and trunk to measure various movements. The 2nd control group completed their measurements and tests at college. Additionally, a clinical test using the American Spinal Injury Association scale (ASIA) was conducted on each participant to assess sensory feeling.
  Interventions: Other: Home-Based Rehabilitation rogram
- First Control Group Five People with SCI (No Intervention): This group only conducted the pre-post1 and post2-tests
- Healthy Group Five people (No Intervention): This group only conducted the pre-post1 and post2-tests

INTERVENTIONS:
Other: Home-Based Rehabilitation rogram — The intervention is distinguished from others in that it applies to patients' homes and the trial was followed up in the middle of complex conditions of the COVID-19 Pandemic. Also, the challenge was represented by the HBRP applied to patients with SCIs after 4-5 years of rehabilitation interruption.
  Other Names: HBRP
  Arms: Rehabilitation program

SUMMARY:
Feasibility of Home-Based Rehabilitation on Body Composition, some Anthropometric Measures and Muscular Strength after interruption 4-5 years of Spinal Cord Injury: Serial Cases Study on ISIS War Survivors in Iraq

Summary Background: The war in Mosul wrecked hospitals and rehab centers, leaving a gap in rehabilitation services. This resulted in a need for alternative solutions for rehabilitation. Objectives: This study aims to create a home-based rehabilitation program (HBRP) that fits the participants' surroundings, and also detect and evaluate how effective it is in improving body composition, some anthropometric measurements, and muscle strength after a (4-5) year break in rehabilitation.

Methods: This voluntary controlled trial included 18 volunteers split into three groups: 13 people with Spinal Cord Injury (SCI) their injuries time since (53.4-55) months. They joined voluntarily into Two groups, Eight in the experimental group (Exp.) and Five in the first control (1st Con.); while Five were healthy individuals in the second control (2nd Con.); all around (21.2) years old on average. The HBRP focused on muscles and whole-body joints by using the basic equipment and exercises right at the patient's homes. The program consisted of five weekly sessions with a gradually increasing achievement time of (45-120) minutes per session, participants were given rest time between exercises based on their level and severity of injury. The assessment was every three months.

DETAILED DESCRIPTION:
Feasibility of Home-Based Rehabilitation on Body Composition, some Anthropometric Measures and Muscular Strength after interruption 4-5 years of Spinal Cord Injury: Serial Cases Study on ISIS War Survivors in Iraq

Summary Background: The war in Mosul wrecked hospitals and rehab centers, leaving a gap in rehabilitation services. This resulted in a need for alternative solutions for rehabilitation. Objectives: This study aims to create a home-based rehabilitation program (HBRP) that fits the participant; surroundings, and also detect and evaluate how effective it is in improving body composition, some anthropometric measurements, and muscle strength after a (4-5) year break in rehabilitation.

Methods: This voluntary controlled trial included 18 volunteers split into three groups: 13 people with Spinal Cord Injury (SCI) their injuries time since (53.4-55) months. They joined voluntarily into Two groups, Eight in the experimental group (Exp.) and Five in the first control (1st Con.); while Five were healthy individuals in the second control (2nd Con.); all around (21.2) years old on average. The HBRP focused on muscles and whole-body joints by using the basic equipment and exercises right at the patient's homes. The program consisted of five weekly sessions with a gradually increasing achievement time of (45-120) minutes per session, participants were given rest time between exercises based on their level and severity of injury. The assessment was every three months.

Innovatively, this study stands out by introducing an HBRP tailored for individuals with SCI after interruption sustained (4 - 5) years ago. This unique approach not only addresses the challenges posed by the interruption of previous rehabilitation efforts but also seeks to uncover the efficacy of rehabilitation in these specific circumstances.

Detailed Description:

Feasibility of Home-Based Rehabilitation on Body Composition, some Anthropometric Measures and Muscular Strength after interruption 4-5 years of Spinal Cord Injury: Serial Cases Study on ISIS War Survivors in Iraq

Background:

Spinal Cord Injury (SCI) is a complex pathology that requires skills in assessment, treatment, and rehabilitation, SCI is a large topic area. Approximately (90%) of SCI cases occur as a result of traumatic causes Globally, incidence varies from 40 to 80 cases per million population. So, people with injuries consequences are becoming more frequent due to conflicts and wars. In Iraq, the main reasons for the occurrence of this injury due to were the Islamic State in Iraq and Syria (ISIS) war, which is resulting in enormous unmet rehabilitation needs. Alarcon Cieza found in his study Rehabilitation the health strategy of the 21st Century that the rehabilitation stakeholders need to bring together the distinct portraits of rehabilitation under the concept of functioning because much of these unmet needs are concentrated amongst the poorest populations in low- and middle-income countries and conflict-affected settings, which are often ill-equipped to cope with these increasing needs for rehabilitation services. Iraq is regarded as one of these countries its health sectors, including rehabilitation, have been exhausted due to wars and armed violence. However, rehabilitation can be effective across almost all conditions, therefore in some ways, we should have been so backwards about recognizing the effectiveness of rehabilitation for many years.

It is worth noting that healthcare problems are among the most complex problems faced by human beings, especially under conditions of war, armed conflicts, terrorist operations and post-war secretions. In low-middle income countries, so many people would die from SCI within a year, two years, or three years from infection, renal failure, and so on, and also people could not work, and they either were at home or in residential care, just waiting to die. One of the defining characteristics of rehabilitation is that there are many interventions; in contrast to most medical conditions, rehabilitation can take place in any setting as a process for problem-solving.

In Iraq, war-related destruction of health institutions and rehabilitation centers has led to a focus on home-based rehabilitation programs (HBRP) and new sporting activities as positive and alternative approaches for rehabilitating individuals with SCI. This article emphasizes the significance of home-based rehabilitation for individuals with SCI to prevent complications that arise from neglecting rehabilitation. Neglecting rehabilitation can result in complex health problems, a major concern observed among the study participants who discontinued rehabilitation due to ineffective and insufficient programs. Additionally, there was a notable mismatch between the participantscircumstances and the available rehabilitation systems and methods. To ensure continuous and successful rehabilitation for individuals with SCI, it is important to implement exercise regimes that intrinsically motivate them. Robert et al, confirmed that rehabilitation can occur at home, and it is a practical matter of what is the best way to organize it so that the patient is safe, the necessary equipment is available, and the therapists and other team members, time is used appropriately. The process is a standard problem-solving process individualized to the patient, which is necessary when solving any problem. Reconsidering rehabilitation at home by introducing new sporting activities has been recognized as a positive and desirable area of rehabilitation 8.

Objectives: Innovatively, this study stands out by introducing an HBRP tailored for individuals with SCI after interruption sustained between (4 - 5) years ago. This unique approach not only addresses the challenges posed by the interruption of previous rehabilitation efforts but also seeks to uncover the efficacy of rehabilitation in these specific circumstances.

The main contributions of this study are:

To the best of the authors' knowledge, this is the first study in Iraq that highlighted the surviving victims of ISIS with SCIs.

The preparation of a home-based rehabilitation program (HBRP) that lasted for six months and that was compatible with the participants' living and environmental conditions as an alternative solution for conditions after the war also, at the time of the COVID-19 pandemic when everything was under the closure.

Assessing the effectiveness of rehabilitation on some anthropometric and physical variables in participants with SCI following participants' stopping of rehabilitation for (4-5) years after SCI.

The study raises two questions Does the home-based rehabilitation program (HBRP) affect people with spinal cord injury through interruption of rehabilitation for 4-5 years? Is the HBRP effects on variables such as body composition (Weight, BMI); Anthropometric Measures, and Muscle strength? Methods: This voluntary controlled trial included 18 volunteers split into three groups: 13 people with Spinal Cord Injury (SCI) their injuries time since (53.4-55) months. They joined voluntarily into Two groups, eight in the experimental group (Exp.) and Five in the first control (1st Con.); while five were healthy individuals in the second control (2nd Con.); all around (21.2) years old on average. As a first procedure, detailed interviews were conducted with each participant at the beginning of the study to gather information about their physical, psychological, and social well-being. This information helped the authors create personalized rehabilitation plans for each participant to ensure their participation in the study for the entire 6 months period. Through our study objectives, the authors used body composition such as height, weight, BMI and some anthropometric measurements for body parts circumferences by using tape measurements, similar to a previous study by Akita et al.. Also, muscle strength tests were performed on participants' lower and upper extremities, head, and trunk to measure various movements. The 2nd control group completed their measurements and tests at college. Additionally, a clinical test using the American Spinal Injury Association scale (ASIA) was conducted on each participant to assess sensory feeling and voluntary movement potential on both sides of the body.

The physical tests were conducted using a handheld muscle tester called MicroFET2 to evaluate the strength of participants' lower extremities, head, and trunk by using unit measure kilogram (kg) 11. The Exp. group underwent a 6-month intensive rehabilitation program that involved whole-body exercises, including stretching, strength, endurance, and aerobic training, which was prepared based on previous studies 12. The program included five weekly sessions of (45-120) minutes, gradually increasing in intensity. It encompassed various exercises like bed exercises, rubber ball exercises for strength and balance, trunk flexibility exercises, crawling, rolling, ball-related movements, and exercises on parallel bars. Also, aerobic exercises targeted cardiorespiratory fitness. While weight exercises focused on the upper limbs, shoulders, chest, and back. Rest periods were personalized based on injury severity and overall health. The authors updated the exercises based on regular assessments every 3 months, tracking muscle strength and endurance. The authors created a contact link for coordination among medical, rehabilitative teams, and participants, families, overcoming some challenges within the Iraqi healthcare system.

To address complex complications like bed sores, renal infections, and muscle atrophy, the authors followed the method of psychological support. This method aimed to stimulate patients, willpower, encouraging them to overcome complications and emphasizing the benefits of rehabilitation for improved overall health and independence, by made WhatsApp group was created to facilitate information sharing and provide visual evidence of successful cases, inspiring and encouraging participants. Furthermore, the participant weight and BMI were monitored due to the potential impact of factors such as limited movement and hormonal changes on weight fluctuations, as recommended in previous studies.

The study highlights the participants the participants fidelity to treatment, as evidenced by positive outcomes and sustained progress beyond the conclusion of the therapeutic experiment. The participants demonstrated loyalty through ongoing communication with the main author, seeking feedback on their rehabilitation stages who reach it. Notably, some participants achieved the significant milestone of walking by standard walker with the assistive device Knee Ankle Foot Orthosis(KAFO).

The study used Two-way ANOVA repeated measures as a statistical analysis method, with effect size and improvement percentage (IP) as measures, and (IBM-SPSS statistics processor version 20) for data analysis. A statistical significance level of P≤ 0.05 (alpha) was used.

ELIGIBILITY:
Inclusion Criteria:

* A spinal cord injury resulting in traumatic injury.
* The participant should have paraplegia and he/she able to use his/her upper limbs to do exercises program

Exclusion Criteria:

* Any person has no traumatic spinal cord injury or his/her injury resulted by such as caused diseases as well as he/she has a tetraplegia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Weight | The period of trial was 6-month. At the beginning before starting the author conducted the pre-tests and after finished 3-month repeated all tests as a post1-test, and at the end of 6-month from the HBRP the author repeated all tests as a post2-test
  It used weight by using the electronic scale if the patient can stand up or can not hold him/her by another person and calculate the weight by subtracting the person's weight from the sum of the weight of both. The unit measure was Kilogram (kg)
Anthropometric Measures (Waist/Abdomen, Pelvis, Both Thigh, Both Legs Circumferences) | The period of trial was 6-month. At the beginning before starting the author conducted the pre-tests and after finished 3-month repeated all tests as a post1-test, and at the end of 6-month from the HBRP the author repeated all tests as a post2-test
  Ii used the tap measure to determine the circumferences of the Abdomen,/waist, Pelvis, Right and Left Thigh, and Right and Left Leg as anthropometric measures. The unit measure was centimeter (cm).
The muscle strength of the lower limbs, head and Trunk | The period of trial was 6-month. At the beginning before starting the author conducted the pre-tests and after finished 3-month repeated all tests as a post1-test, and at the end of 6-month from the HBRP the author repeated all tests as a post2-test
  The physical tests were conducted using a handheld muscle tester called MicroFET2 to evaluate the strength of participants' lower extremities, head, and trunk by using unit measure kilogram (kg) from positions (lying-down, supine, on the ground and in the bed)
Body mass index (BMI) | The period of trial was 6-month. At the beginning before starting the author conducted the pre-tests and after finished 3-month repeated all tests as a post1-test, and at the end of 6-month from the HBRP the author repeated all tests as a post2-test
  It used the criteria of BMI according to WHO

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sfax, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
The authors agree to share the data of study after the study will be published online and after a request by email
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study published online for 10 months
Access Criteria: Any author needs the data or information about the study methods, he/she will be able to get it by contact with following this email and phone:
  m.a.fathi@uomosul.edu.iq 009647701680770
URL: https://uomosul.edu.iq/?fbclid=IwAR1UpByF7HKCbKITGt3xlTSObKzfkVs_aFuWy2WBVPc10wa9OjxaiL5rouI

REFERENCES:
- [Background] Duran FS, Lugo L, Ramirez L, Eusse E. Effects of an exercise program on the rehabilitation of patients with spinal cord injury. Arch Phys Med Rehabil. 2001 Oct;82(10):1349-54. doi: 10.1053/apmr.2001.26066. PMID 11588736
- [Background] Abilmona SM, Sumrell RM, Gill RS, Adler RA, Gorgey AS. Serum testosterone levels may influence body composition and cardiometabolic health in men with spinal cord injury. Spinal Cord. 2019 Mar;57(3):229-239. doi: 10.1038/s41393-018-0207-7. Epub 2018 Oct 22. PMID 30349112
- [Background] Khorasanizadeh M, Yousefifard M, Eskian M, Lu Y, Chalangari M, Harrop JS, Jazayeri SB, Seyedpour S, Khodaei B, Hosseini M, Rahimi-Movaghar V. Neurological recovery following traumatic spinal cord injury: a systematic review and meta-analysis. J Neurosurg Spine. 2019 Feb 15;30(5):683-699. doi: 10.3171/2018.10.SPINE18802. Print 2019 May 1. PMID 30771786
- [Result] Modlesky CM, Bickel CS, Slade JM, Meyer RA, Cureton KJ, Dudley GA. Assessment of skeletal muscle mass in men with spinal cord injury using dual-energy X-ray absorptiometry and magnetic resonance imaging. J Appl Physiol (1985). 2004 Feb;96(2):561-5. doi: 10.1152/japplphysiol.00207.2003. Epub 2003 Oct 3. PMID 14527962
- [Result] Gorgey AS, Dolbow DR, Dolbow JD, Khalil RK, Gater DR. The effects of electrical stimulation on body composition and metabolic profile after spinal cord injury--Part II. J Spinal Cord Med. 2015 Jan;38(1):23-37. doi: 10.1179/2045772314Y.0000000244. Epub 2014 Jul 8. PMID 25001669
- [Result] Yuen J, Thiyagarajan CA, Belci M. Patient experience survey in telemedicine for spinal cord injury patients. Spinal Cord. 2015 Apr;53(4):320-3. doi: 10.1038/sc.2014.247. Epub 2015 Jan 27. PMID 25622730
- [Result] Richard-Denis A, Dionne A, Mputu PM, Mac-Thiong JM. Do all patients with functional motor-incomplete (AIS-D) traumatic spinal cord injury need specialized inpatient functional rehabilitation? A prospective observational cohort study proposing clinical criteria for home-based rehabilitation after acute care. J Spinal Cord Med. Published online 2023. doi:10.1080/10790268.2023.2200354 25. Hicks AL, Martin KA, Ditor DS, et al. Long-term exercise training in persons with spinal cord injury: Effects on strength, arm ergometry performance and psychological well-being. Spinal Cord. 2003;41(1):34-43. doi:10.1038/sj.sc.3101389
- [Result] Hicks AL, Martin KA, Ditor DS, Latimer AE, Craven C, Bugaresti J, McCartney N. Long-term exercise training in persons with spinal cord injury: effects on strength, arm ergometry performance and psychological well-being. Spinal Cord. 2003 Jan;41(1):34-43. doi: 10.1038/sj.sc.3101389. PMID 12494319
- [Result] Richard-Denis A, Dionne A, Mputu PM, Mac-Thiong JM. Do all patients with functional motor-incomplete (AIS-D) traumatic spinal cord injury need specialized inpatient functional rehabilitation? A prospective observational cohort study proposing clinical criteria for home-based rehabilitation after acute care. J Spinal Cord Med. 2024 Sep;47(5):753-764. doi: 10.1080/10790268.2023.2200354. Epub 2023 Apr 21. PMID 37083554
- [Result] Ji X, Xu Z, Liu D, Chen Y. Effects of exercise training on neurological recovery, TGF-beta1, HIF-1alpha, and Nogo-NgR signaling pathways after spinal cord injury in rats. Clinics (Sao Paulo). 2023 Jul 27;78:100236. doi: 10.1016/j.clinsp.2023.100236. eCollection 2023. PMID 37515927
- See also: This scientific association aims to develop the members and participant in rehabilitation — https://members.physio-pedia.com/learn/
- See also: The CSRO is dedicated to the funding of targeted research to maximize functional recovery and cure paralysis caused by spinal cord injury. We envision a world without paralysis caused by spinal cord injury. — https://sci-can.ca/network

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: study protocol included the statistically analysis (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT06230627/Prot_SAP_001.pdf
  • Study Protocol: Proposal of study (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT06230627/Prot_002.pdf
  • Informed Consent Form: Decision of Committee of Ethical Approval (2021-11-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT06230627/ICF_003.pdf
  • Informed Consent Form: locally Ethical Approval (2021-07-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT06230627/ICF_004.pdf